CLINICAL TRIAL: NCT02920567
Title: Impact of Prophylactic Octreotide to Pancreatic Exocrine Secretion and Pancreatic Fistula After Pancreatoduodenectomy
Brief Title: Impact of Prophylactic Octreotide to Pancreatic Exocrine Secretion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saint Vincent's Hospital, Korea (Other)
Responsible Party: Principal Investigator, YOU DONG DO, Associated Professor, Saint Vincent's Hospital, Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XC12MIMI0138V
Record Dates: First submitted 2016-09-28; First posted 2016-09-30 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Periampullary Tumors
MeSH Terms: interventions — Octreotide; Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- octreotide (Experimental): After pancreatoduodenectomy, octreotide was injected to patients every 8 hours subcutaneously for 7 days
  Interventions: Drug: Octreotide
- Placebo (Placebo Comparator): After pancreatoduodenectomy, normal saline was injected to patients every 8 hours subcutaneously for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Octreotide — After pancreatoduodenectomy, octreotide was injected to patients every 8 hours subcutaneously for 7 days
  Other Names: Treatment
  Arms: octreotide
Drug: Placebo — After pancreatoduodenectomy, normal saline was injected to patients every 8 hours subcutaneously for 7 days
  Other Names: control
  Arms: Placebo

SUMMARY:
This study aims to examine whether octreotide has an effect on inhibition of the exocrine secretion fo the pancreas, which might lower the rate of postoperative pancreatic fistula after pancreatoduodenectomy. Patients who will undergo pancreatoduodenectomy for periampullary tumors were enrolled. The patients were randomly assigned to intervention (use of octreotide) or placebo groups. Octreotide was injected subcutaneously every 8 hours for 7 days. Every patients will undergo pancreaticojejunostomy with external stent for remnant pancreas management. The pancreatic juice is drained through the external stent by negative pressure and amounted.

Primary endpoint was the amount of pancreatic juice for each postoperative day. Secondary endpoint was the rate of pancreatic fistula.

DETAILED DESCRIPTION:
This study aims to examine whether octreotide has an effect on inhibition of the exocrine secretion fo the pancreas, which might lower the rate of postoperative pancreatic fistula after pancreatoduodenectomy. Patients who will undergo pancreatoduodenectomy for periampullary tumors were enrolled. The patients were randomly assigned to intervention (use of octreotide) or placebo groups. Octreotide of 100ug(1mL) was injected subcutaneously just before operation and every 8 hours for 7 days postoperatively. The placebo group was managed with normal saline (1mL) for same period. Every patients will undergo pancreaticojejunostomy with external stent for remnant pancreas management. The pancreatic juice is drained through the external stent by negative pressure (Barovac) and amounted.

Postoperative care of patients was same between groups such as pain control and supportive care. The amount of drained pancreatic juice via external stent was recorded everyday.

Primary endpoint was the amount of pancreatic juice for each postoperative day. Secondary endpoint was the rate of pancreatic fistula.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo pancreatoduodenectomy for periampullary tumors

Exclusion Criteria:

* Patients with preoperative pancreatitis
* Patients who did not undergo pancreatoduodenectomy
* Patients who underwent bypass surgery or total pancreatectomy
* Patients who injection of octreotide less than 5 days

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2014-01; Primary Completion 2018-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Amount of pancreatic secretion | 1 day

SECONDARY OUTCOMES:
Rate of pancreatic fistula | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Dong Do You, MD, PhD, Study Director — The Catholic University of Korea
Locations (1):
- the Catholic University of Korea St. Vincent's Hospital, Suwon, South Korea

REFERENCES:
- [Background] Bauer W, Briner U, Doepfner W, Haller R, Huguenin R, Marbach P, Petcher TJ, Pless. SMS 201-995: a very potent and selective octapeptide analogue of somatostatin with prolonged action. Life Sci. 1982 Sep 13;31(11):1133-40. doi: 10.1016/0024-3205(82)90087-x. PMID 6128648
- [Background] Buchler M, Friess H, Klempa I, Hermanek P, Sulkowski U, Becker H, Schafmayer A, Baca I, Lorenz D, Meister R, et al. Role of octreotide in the prevention of postoperative complications following pancreatic resection. Am J Surg. 1992 Jan;163(1):125-30; discussion 130-1. doi: 10.1016/0002-9610(92)90264-r. PMID 1733360
- [Background] Di Carlo V, Chiesa R, Pontiroli AE, Carlucci M, Staudacher C, Zerbi A, Cristallo M, Braga M, Pozza G. Pancreatoduodenectomy with occlusion of the residual stump by Neoprene injection. World J Surg. 1989 Jan-Feb;13(1):105-10; discussion 110-1. doi: 10.1007/BF01671167. PMID 2543144